CLINICAL TRIAL: NCT05297695
Title: Effect of Treating Helicobacter Pylori Infection on Seizure Frequency in Children With Drug-Resistant Idiopathic Generalized Epilepsy
Brief Title: Helicobacter Pylori Eradication Therapy for Epileptic Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mena Samy Basily, Principal Investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: soh-med-22-03-13
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Epilepsy, Generalized; Helicobacter Pylori Infection
Keywords: Children; Epilepsy; Helicobacter pylori; Treatment; Seizure
MeSH Terms: conditions — Epilepsy, Generalized; Epilepsy; Seizures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Children with drug-resistant idiopathic generalized epilepsy and positive H. pylori stool antigen test who will receive H. pylori eradication therapy.
  Interventions: Drug: Triple therapy for H. pylori infection
- Control group (No Intervention): Children with drug-resistant idiopathic generalized epilepsy and positive H. pylori stool antigen test who will not receive H. pylori eradication therapy.

INTERVENTIONS:
Drug: Triple therapy for H. pylori infection — Triple therapy for H. pylori infection (Esomeprazole, Amoxicillin, and Clarithromycin) for two weeks
  Arms: Study group

SUMMARY:
Helicobacter pylori (H. pylori) infection is associated with several health problems. The role of H. pylori infection in epilepsy has been investigated in a few studies. To the best of our knowledge, there have been no previous studies on the effect of treating H. pylori infection on seizure frequency among children with drug-resistant idiopathic generalized epilepsy. This study aims to evaluate the effect of treating H. pylori infection on seizure frequency among children with drug-resistant idiopathic generalized epilepsy.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) is a spiral-shaped Gram-negative bacterium, which causes chronic infection in more than 50% of human population. H. pylori infection is associated with several gastrointestinal disorders, such as gastritis and gastric/duodenal ulcers. Moreover, accumulating body of evidence indicates the possible role of H. Pylori infection in extraintestinal health problems, such as iron deficiency anemia, immune thrombocytopenic purpura (ITP), numerous dermatological diseases, Alzheimer disease, Parkinson's disease, multiple sclerosis, and epilepsy.

Epilepsy is a common neurological disorder characterized by recurrent unprovoked seizures. This condition affects 0.5% to 1% of all children and is associated with neurobiological, cognitive, psychological, and social consequences. Seizures can usually be controlled by anti-epileptic drugs (AEDs) in up to two-thirds of children with epilepsy. However, this leaves a significant part of epileptic children whose seizures are not controlled by pharmacotherapy.

The development of epilepsy is highly complex and can be attributed to multiple etiologies classified into structural (e.g., malformation, trauma, ischemia), genetic, infectious, metabolic, and immune factors. However, the etiology remains unknown in about half of epileptic children. Idiopathic generalized epilepsies (IGE) constitute about one-third of all epilepsies. Efforts to explore new possible mechanisms contributing to the development of epilepsy, particularly drug-resistant IGE, could contribute to the development of new therapeutic strategies to improve patients' outcomes.

The role of H. pylori infection in epilepsy has been investigated in a few studies, some of which reported that the seroprevalence of H. pylori infection is significantly higher in patients with idiopathic epilepsy compared with patients with other chronic diseases, and that H. pylori infection is associated with poor prognosis.

Potential H. pylori-induced epileptic effects are probably immune-mediated that can be attributed to a cross-mimicry mechanism between H. pylori and human cellular phospholipids with production of autoimmune antibodies (e.g., anti-cardiolipin) and H. pylori infection-related activation of pro-inflammatory cells with systemic release of proinflammatory cytokines (e.g., IL-6, 8 and TNF- α) which are involved in disruption of the blood-brain barrier and neuroinflammation.

To the best of our knowledge, there have been no previous studies on the effect of treating H. pylori infection on seizure frequency among children with drug-resistant IGE. This study aims to evaluate the effect of treating H. pylori infection on seizure frequency among children with drug-resistant IGE.

ELIGIBILITY:
Inclusion Criteria:

* Age between 4 and 18 years.
* Idiopathic generalized epilepsies (IGE), including childhood absence epilepsy, juvenile absence epilepsy, juvenile myoclonic epilepsy, or IGE with generalized tonic-clonic seizures only (IGE-TCS).
* Drug-resistant epilepsy, defined as failure of adequate trials of two tolerated and appropriately chosen and used anti-epileptic drugs schedules (whether as monotherapies or in combination) to achieve sustained seizure freedom
* Positive H. pylori stool antigen (HpSA) test (at initial screening).

Exclusion Criteria:

* Failure to obtain informed consent.
* Presence of a medical indication for treating H. pylori infection, including gastric or duodenal ulcer, chronic immune thrombocytopenic purpura, and refractory iron deficiency anemia.
* Known allergy or contraindications to any of the study drugs.
* Treatment with antibiotics and/or proton pump inhibitors in the last 2 months.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Seizure improvement | 2.5 months following H. pylori eradication therapy
  ≥ 50% seizure frequency reduction compared with baseline

SECONDARY OUTCOMES:
Need for escalation of antiepileptic drugs | 2.5 months following H. pylori eradication therapy
  Need for escalation of antiepileptic drugs compared with baseline
Occurrence of status epilepticus | 2.5 months following H. pylori eradication therapy
Occurrence of adverse effects of H. pylori eradication therapy | 2.5 months following H. pylori eradication therapy

CONTACTS AND LOCATIONS:
Overall Officials: Montaser M Mohamed, MD, PhD, Study Chair — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the study
Access Criteria: Data will be available for researchers upon reasonable request

REFERENCES:
- [Background] Korotkaya Y, Shores D. Helicobacter pylori in Pediatric Patients. Pediatr Rev. 2020 Nov;41(11):585-592. doi: 10.1542/pir.2019-0048. PMID 33139411
- [Background] Fine A, Wirrell EC. Seizures in Children. Pediatr Rev. 2020 Jul;41(7):321-347. doi: 10.1542/pir.2019-0134. PMID 32611798
- [Background] Scheffer IE, Berkovic S, Capovilla G, Connolly MB, French J, Guilhoto L, Hirsch E, Jain S, Mathern GW, Moshe SL, Nordli DR, Perucca E, Tomson T, Wiebe S, Zhang YH, Zuberi SM. ILAE classification of the epilepsies: Position paper of the ILAE Commission for Classification and Terminology. Epilepsia. 2017 Apr;58(4):512-521. doi: 10.1111/epi.13709. Epub 2017 Mar 8. PMID 28276062
- [Background] Fisher RS, Acevedo C, Arzimanoglou A, Bogacz A, Cross JH, Elger CE, Engel J Jr, Forsgren L, French JA, Glynn M, Hesdorffer DC, Lee BI, Mathern GW, Moshe SL, Perucca E, Scheffer IE, Tomson T, Watanabe M, Wiebe S. ILAE official report: a practical clinical definition of epilepsy. Epilepsia. 2014 Apr;55(4):475-82. doi: 10.1111/epi.12550. Epub 2014 Apr 14. PMID 24730690
- [Background] Yao G, Wang P, Luo XD, Yu TM, Harris RA, Zhang XM. Meta-analysis of association between Helicobacter pylori infection and multiple sclerosis. Neurosci Lett. 2016 May 4;620:1-7. doi: 10.1016/j.neulet.2016.03.037. Epub 2016 Mar 23. PMID 27033666
- [Background] Okuda M, Miyashiro E, Nakazawa T, Minami K, Koike M. Helicobacter pylori infection and idiopathic epilepsy. Am J Med. 2004 Feb 1;116(3):209-10. doi: 10.1016/j.amjmed.2003.05.005. No abstract available. PMID 14749171
- [Background] Ozturk A, Ozturk CE, Ozdemirli B, Yucel M, Bahcebasi T. Helicobacter pylori infection in epileptic patients. Seizure. 2007 Mar;16(2):147-52. doi: 10.1016/j.seizure.2006.10.015. Epub 2006 Nov 27. PMID 17126040
- [Background] Kwan P, Arzimanoglou A, Berg AT, Brodie MJ, Allen Hauser W, Mathern G, Moshe SL, Perucca E, Wiebe S, French J. Definition of drug resistant epilepsy: consensus proposal by the ad hoc Task Force of the ILAE Commission on Therapeutic Strategies. Epilepsia. 2010 Jun;51(6):1069-77. doi: 10.1111/j.1528-1167.2009.02397.x. Epub 2009 Nov 3. PMID 19889013
- [Derived] Mohamed MA, Mahmoud EA, Basily MS, Mohamed MM, Ahmed OAA, Abdelkreem E. Efficacy of treating Helicobacter pylori infection on seizure frequency in children with drug-resistant idiopathic generalized epilepsy: a randomized controlled trial. Ital J Pediatr. 2025 Apr 17;51(1):121. doi: 10.1186/s13052-025-01956-2. PMID 40247384